CLINICAL TRIAL: NCT03614806
Title: Transcutaneous Carbon Dioxide Pressure (tcPCO2) Monitoring Vs End-tidal Partial Pressure Carbon Dioxide (PetCO2) Measurement in the Diagnosis of Hyperventilation Syndrome (HVS) (TCvsPETCO2 )
Brief Title: Comparison of Transcutaneous Vs End-tidal CO2 Pressure Measurements in Hyperventilation Syndrome Diagnosis
Acronym: TCvsPETCO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/128/HP
Record Dates: First submitted 2017-11-29; First posted 2018-08-03 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Hyperventilation Syndrome; Hypocapnia; Alkalosis, Respiratory; Hyperventilation
MeSH Terms: conditions — Hypocapnia; Alkalosis, Respiratory; Hyperventilation

STUDY DESIGN:
Intervention Model Description: open label study prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients tested for hyperventilation (Experimental): Simultaneous Transcutaneous and End-tidal CO2 measurements. Eligible patients will be first invited to fill in the Nijmegen questionnaire. Then, in an hyperventilation test, transcutaneous Carbon Dioxide Pressure will be recorded simultaneously with the standard End-tidal Carbon Dioxide Pressure measurement.
  Interventions: Diagnostic Test: Simultaneous Transcutaneous and End-tidal CO2 measurements

INTERVENTIONS:
Diagnostic Test: Simultaneous Transcutaneous and End-tidal CO2 measurements — Included patients will be invited to fill in the Nijmegen questionnaire. During the hyperventilation test, PtcCO2 (mmHg) will be recorded simultaneously with the standard End-tidal Cpartial pressure CO2 measurement

SUMMARY:
Hyper Ventilation Syndrome is a frequent disease affecting adults whose diagnosis is often belated or even unrecognized due to the lack of "gold standard" criteria. Its diagnosis currently relies on the Nijmegen score associated with a PetCO2 assesment using a hyperventilation provocation test. Correlation between Nijmegen Questionnaire scores and PetCO2 appears highly variable. PtcCO2 monitoring is a noninvasive alternative method providing a continuous estimation of arterial CO2 pressure (PaCO2) which could represent an advantageous alternative to PetCO2 measurements. Several reports have demonstrated that PtcCO2 monitoring reflects more faithfully PaCO2 than PetCO2, no study have evaluated its value in this indication.

The primary aim of the study is to compare the diagnostic value of PtcPCO2 monitoring with PetCO2, the method currently used.

Included patient will be invited to fill in the Nijmegen questionnaire and an ambient air gas measurement will be performed. PtcCO2 (mmHg) will be simultaneously measured during hyperventilation test. Nijmegen score signs reproduced by the test will be analysed. HVS diagnosis will be assessed by usual criteria (PetCO2 <30 mmHg at the end of hyperventilation test or under the PetCO2 value at rest, Nijmegen score> 23).

PtcCO2 data will be blinded interpreted later. We will compare if PetCO2 and PtcCO2 leads to the same diagnosis or not.

DETAILED DESCRIPTION:
Primary Goal:

Show that the use of either of the two pCO2 measurements leads to the same diagnostic conclusion in HVS diagnosis with a likelihood greater than 80 %.

Secondary Outcome Measures :

Evaluate the correlation between PtcCO2 and PtcCO2 measurements Evaluate tolerance to the hyperventilation test

Inclusion Criteria :

1. The patient must have reached the age of the civil majority (≥ 18 yo)
2. All patients refered to the Physiology department of Rouen University Hospital, France, for an hyperventilation test
3. The patient must be a member or beneficiary of a health insurance program
4. The patient must have given his / her free and informed consent and signed the consent

Exclusion Criteria :

1. Sepsis
2. Hypercapnia (PaCO2 > 50mmHg)
3. Patient treated by long-term oxygen therapy
4. Subjects under judicial protection, or adults under any kind of guardianship or under judicial control
5. Pregnancy or breastfeeding women
6. Electrolytic unbalance
7. Hyperthyroidism
8. Neurological disease
9. Probability of drug-induced hyperventilation (progestagens , aspirin, beta agonists)

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have reached the age of the civil majority (≥ 18 yo)
2. All patients refered to the Physiology department of Rouen University Hospital, France, for an hyperventilation test
3. The patient must be a member or beneficiary of a health insurance program
4. The patient must have given his / her free and informed consent and signed the consent

Exclusion Criteria:

1. Sepsis
2. Hypercapnia (PaCO2 > 50mmHg)
3. Patient treated by long-term oxygen therapy
4. Subjects under judicial protection, or adults under any kind of guardianship or under judicial control
5. Pregnancy or breastfeeding women
6. Electrolytic unbalance
7. Hyperthyroidism
8. Neurological disease
9. Probability of drug-induced hyperventilation (progestagens , aspirin, beta agonists)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Trans-cutaneous Carbon Dioxide pressure | during hyperventilation test
  Trans-cutaneous Carbon Dioxide pressure measurements diagnostic of hyperventilation syndrome will be evaluated by comparing it with that of standard
End-tidal Carbon Dioxide partial pressure | during hyperventilation test
  End-tidal Carbon Dioxide partial pressure measurement. Consistency of the diagnostic conclusions reached by either test will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: ARTAUD-MACARI Elise, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Physiology department of Rouen University Hospital,, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided